CLINICAL TRIAL: NCT04366115
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study Evaluating AVM0703 in Patients With Acute Respiratory Distress Syndrome
Brief Title: Evaluating AVM0703 for Treatment of COVID-19 or Influenza-mediated ARDS
Acronym: AVM0703
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AVM Biotechnology Inc (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVM0703-101
Record Dates: First submitted 2020-04-26; First posted 2020-04-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: ARDS; Covid19; Influenza, Human
Keywords: ARDS; COVID19; Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Intervention Model Description: This is a two-armed randomized, double-blinded, placebo control controlled study. Each arm (one arm of COVID-19 mediated ARDS and one arm of influenza (A or B) mediated ARDS will be randomized to 3:1 (active to placebo)
Who Masked: Participant, Care Provider, Investigator
Masking Description: The pharmacist will prepare the infusion solution and medication for delivery to the patient's bedside for administration. The active and placebo medications look identical, preventing care-givers and the participant from breaking the blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- AVM0703 COVID-19 ARDS - active (Active Comparator): Supra-pharmacologic dexamethasone sodium phosphate
  Interventions: Drug: AVM0703
- Placebo COVID-19 ARDS - placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo
- AVM0703 Influenza ARDS - active (Active Comparator): Supra-pharmacologic dexamethasone sodium phosphate
  Interventions: Drug: AVM0703
- AVM0703 Influenza ARDS - placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVM0703 — Single IV infusion at 10 mg/mL in normal saline over 1 hour to patients.
  Other Names: Suprapharmacologic dexamethasone sodium phosphate
  Arms: AVM0703 COVID-19 ARDS - active; AVM0703 Influenza ARDS - active
Drug: Placebo — Single IV infusion in normal saline over 1 hour to patients.
  Arms: AVM0703 Influenza ARDS - placebo; Placebo COVID-19 ARDS - placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled study of AVM0703 administered as a single intravenous (IV) infusion to patients with moderate or severe immediately life-threatening Acute Respiratory Distress Syndrome (ARDS) due to COVID-19 or influenza (A or B). The study is designed to evaluate the safety, tolerability, and pharmacokinetics of single dose of AVM0703 in these ARDS patients.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety and tolerability of a single dose of AVM0703 in patients with moderate, severe or immediately life-threatening ARDS due to COVID-19 or Influenza (A or B) infection.

The secondary objectives of the study are to 1) evaluate the pharmacokinetics (PK) and 2) evaluate potential clinical findings following a single dose of AVM0703.

The exploratory objective of the study is to assess potential biomarkers indicative of natural killer T (NKT) cell activity and biomarkers predictive of response to AVM0703 in peripheral blood and bronchoalveolar lavage.

The results of the Phase 1 study will guide the design of the Phase 2 study.

ELIGIBILITY:
Inclusion Criteria

Patients who meet all of the following criteria will be eligible to participate in the study:

1. Age ≥18 years;
2. Must have laboratory confirmed COVID-19;
3. Must have moderate or severe, immediately life-threatening COVID-19 or Influenza (A or B), as follows:

   a. COVID-19 patients with ARDS (Berlin Criteria) as demonstrated by:

   i. Chest radiograph or CT scan showing bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules;

   ii. Respiratory failure not fully explained by cardiac failure or fluid overload; and

   iii. Impaired oxygenation defined as Moderate (partial pressure of oxygen [PaO2]:fraction of inspired oxygen [FiO2] ratio 100 mm Hg to <200 mm Hg with positive end-expiratory airway pressure [PEEP] >5 cm H2O) or Severe (PaO2:FiO2 ratio <100 mm Hg with PEEP>5 cm H2O) on more than 2 arterial blood gases at least 6 hours apart within a 24 hour period;

   b. Influenza (A or B) patients with ARDS (Berlin Criteria) as demonstrated by:

   i. Chest radiograph or CT scan showing bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules;

   ii. Respiratory failure not fully explained by cardiac failure or fluid overload; and

   iii. Impaired oxygenation defined as Severe (PaO2:FiO2 ratio<100 mm Hg with PEEP >5 cm H2O) on more than 2 arterial blood gases at least 6 hours apart within a 24 hour period;
4. Requires invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) despite standard of care rescue measures (eg, prone positioning, and/or PEEP ladder, and/or inhaled pulmonary vasodilators, and/or recruitment maneuvers and/or neuromuscular blockade);
5. Females of childbearing potential must have a negative serum pregnancy test at screening;
6. Females of childbearing potential and nonsterile males must agree to use medically effective methods of contraception from the time of informed consent through 1 month after study drug infusion; and
7. Capable of providing informed consent, or if not capable, a legally authorized representative is capable of providing informed consent

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from participation in the study:

1. Moribund patient who, in the opinion of the Investigator, is not expected to survive at least 24 hours;
2. Known hypersensitivity or allergy to the study drug or any of its excipients;
3. D-dimer level >3 times above normal range;
4. Known gastric or duodenal ulcer;
5. Uncontrolled type 1 or type 2 diabetes, per judgment of the Investigator;
6. Active and untreated bacterial, fungal, parasitic, or viral infection other than COVID-19 or Influenza (A or B). Patients with a history of a positive hepatitis B surface antigen and/or hepatitis B core antibody must have a negative hepatitis B polymerase chain reaction (PCR) assay result. Patients with history of a positive hepatitis C virus antibody test must have a negative hepatitis C PCR assay result;
7. Positive testing for tuberculosis during screening;
8. Known to have received a live vaccine within the previous 1 month;
9. Immunocompromised patients, defined as those who have received a bone marrow or solid organ transplant on immunosuppressive therapy; or history of human immunodeficiency virus (HIV) infection who have not been taking anti retroviral therapy for at least 6 months before enrollment and/or with most recent CD4 count <200 cells/mL and/or most recent detectable viral load within the previous 6 months;
10. Moderate to End-stage liver disease (Childs-Pugh Score >10);
11. Dialysis-dependent due to underlying chronic renal disease. Note: patients who require dialysis for treatment of renal failure due to complications of COVID-19 or Influenza (A or B) infection are not excluded from enrollment;
12. Significant cardiovascular disease (eg, myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 3 months prior to the start of AVM0703 administration, including: angina requiring therapy, symptomatic peripheral vascular disease, New York Heart Association Class III or IV congestive heart failure, left ventricular ejection fraction <30%, left ventricular fractional shortening <20%, or uncontrolled Grade 3 hypertension (diastolic blood pressure [DBP] >100 mm Hg or systolic blood pressure [SBP] >150 mm Hg) despite antihypertensive therapy.

    Note: patients with heart failure requiring medical support due solely to complications of COVID-19 infection are not excluded from enrollment;
13. Significant screening 12-lead ECG abnormalities, including unstable cardiac arrhythmia requiring medication, atrial fibrillation/flutter, left bundle-branch block, second degree atrioventricular (AV) block type 2, third-degree AV block, Grade 2 bradycardia, or heart rate corrected QT interval using Fridericia's formula average of triplicate ECGs >450 ms;
14. Manic-depressive disorder, schizophrenia, or a history of severe depression or substance abuse;
15. Pregnant or breastfeeding;
16. Concurrent enrollment in any other clinical study involving administration of a novel (ie, unapproved or not considered standard of care) investigational pharmacological agent(s). Concurrent enrollment in observational and device studies and studies involving administration of pharmacological agent(s) approved for other indications or considered emerging standard of care for treatment of COVID-19 (eg, hydroxychloroquine, remdesivir, low-dose dexamethasone), will be allowed if approved by the Sponsor;
17. Treatment with standard of care or off-label treatments for COVID-19 (eg, remdesivir), not administered as part of a formal clinical study, where the first dose was initiated within 72 hours of study drug start; and
18. Inability to obtain informed consent from the patient or legally authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2031-12-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities | 0-12 months
  The primary endpoint of the Phase 1 portion of the study is to evaluate the safety of AVM0703 in subjects with severe or life-threatening COVID-19 infection, and to identify the RP2D.
28 day all-cause mortality will be a primary end point for Phase 1 and 2 | 0-12 months
  The primary endpoint of the Phase 1/2 portion of the study is to evaluate the efficacy of AVM0703 in subjects with severe or life-threatening COVID-19 infection.

IPD SHARING:
Plan to Share IPD: No